CLINICAL TRIAL: NCT06180915
Title: The Effect of Peer Education Based on Assertiveness Skills on Dating Violence Attitudes and Internalized Misogyny
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gazi University (Other)
Collaborators: Tarsus University (Other); Mersin University (Other)
Responsible Party: Principal Investigator, Şengül Yaman Sözbir, Professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: bsrgk33
Record Dates: First submitted 2023-10-30; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Dating Violence
Keywords: dating violence; İnternalized misogyny

STUDY DESIGN:
Intervention Model Description: In order to ensure similarity between groups; Stratified block randomization will be used to assign the women in the sample group to the experimental and control groups. According to the stratified block randomization method, imbalances that may arise in the experimental and control groups are limited. In this method, after stratification according to risk factors, block randomization is performed within each stratum (Akın & Koçoğlu, 2017; Kanık, Taşdelen & Erdoğan, 2011). 1st Layer: 1st grade students. 2nd Layer: 2nd grade students. 3rd Layer: 3rd Grade. grade students In order to determine which stratum group the woman who is found to meet the research criteria and agrees to participate in the study is in, blocks will be created with a combination of 8 and an assignment list will be determined through the website www.randomizer.org.
  Mersin and Tarsus University Midwifery departments were chosen due to the similarity of their core curricula and education in similar geography.
Who Masked: Participant, Outcomes Assessor
Masking Description: Stratified block randomization will be used to prevent selection bias. In this study regarding application bias, it was ensured that the researcher and the participants had not met before and that the researcher did not play a direct role in the academic success of the participants. Researcher and participant blinding will not be possible. Because the researcher will perform the application himself and placebo will not be used in the intervention.
  Pretest and posttests to prevent detection bias will be administered online via Google Forms®, independently of the researcher.
  To prevent reporting bias, the data obtained from the research will be coded as A and B by an independent researcher and transferred to the SPSS program. Analysis of the data will also be done by an independent statistician.
  In order to prevent attrition bias, Attrition Bias and Intention to Treat Test will be used in case of attrition/reduction in the sample group or if the final tests are not completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants will be informed that they must answer the surveys and forms completely and appropriately, as well as attend all training sessions and fulfill their session duties. At the end of the 3-week training program (interim measurement) and 4 weeks later (post-test), the Rathus Assertiveness Inventory, Internalized Misogyny Scale and Flirting Violence Attitude Scale will be converted into an online survey via Google Forms®, the link will be sent to the participants and they will be asked to fill it out.
  Interventions: Behavioral: The peer trainer will be subjected to assertiveness training based on dating violence and internalized misogyny by the researcher for 2 hours a day for 5 days.
- Control Group (No Intervention): The control group will not be subjected to any training. The Control Group will fill out the Introductory Information Form, Rathus Assertiveness Inventory, Internalized Misogyny Scale, Flirting Violence Scale and Cyber Flirting Violence Scale simultaneously with the experimental group at the beginning of the study.

INTERVENTIONS:
Behavioral: The peer trainer will be subjected to assertiveness training based on dating violence and internalized misogyny by the researcher for 2 hours a day for 5 days. — The peer trainer will be subjected to assertiveness training based on dating violence and internalized misogyny by the researcher for 2 hours a day for 5 days. The peer educator will create a Whatsapp group with the experimental group participants and a name for the group will be found by mutual decision. The peer educator will schedule a time and date with the group. Each session will last approximately 60 minutes and the total training duration will be planned to be 3 weeks. One week and one month after the training is completed, the participants will fill out the scales again.
  Arms: Experimental Group

SUMMARY:
This study will be conducted to evaluate the effect of assertiveness training given through peer education on dating violence attitudes and internalized misogyny. In this study ; Nursing takes a role in helping individuals obtain and protect their rights as part of its advocacy role, investigates the obstacles to assertive behavior and solutions to develop assertive behavior as part of its researcher role, takes a role in educating individuals on assertiveness as part of its educational role, and finds solutions to individuals' problems as part of its consultancy role. It will play an active role in students' roles such as being able to produce, providing problem-solving skills with appropriate coping methods.

This study aims to empower women by providing a positive change in the perception of dating violence attitudes and internalized misogyny through peer education based on assertiveness training. It is thought that with this study, the assertiveness behavior of female students studying at the university will be improved and a positive change will be achieved in the perception of dating violence attitudes and internalized misogyny.

The population of the study is female students studying at the university, and female students studying in the midwifery department were selected due to the high density of female students. Female students of Tarsus University Midwifery Department were selected as the intervention group and female students of Mersin University were selected as the control group.

DETAILED DESCRIPTION:
One of the most important problems caused by gender inequality is violence against women. Violence against women is the intimidation of women by using physical force or intimidation, and it covers a wide range of harmful behaviors directed at women and girls because of their gender. The inequality experienced by women regarding their participation in education, paid workforce and decision-making mechanisms negatively affects their access to economic and social resources. Any physical, verbal, psychological, sexual violence and maltreatment that occurs within a dating relationship is considered dating violence. Dating violence negatively affects the individual's quality of life by causing negative effects on a person's self-confidence and self-esteem. Adolescence is a period in which the individual develops an identity, is more questioning, reactive, sensitive, fragile and inexperienced towards life, society and norms compared to other developmental periods, and adopts the values of peer groups. Considering that dating relationships are generally established in adolescence and youth, lack of experience at a young age is one of the effective risk factors for this type of violence. Studies have shown that individuals who experience dating violence during the adolescence period, when vital values are newly formed, have no awareness of the violence experienced, or even if they have awareness, they cannot find a solution to this problem. Exposure to dating violence during adolescence chronicizes the violence, increasing the risk of being both a victim of violence and a perpetrator of violence in adulthood. Women, who have a more passive role due to their gender roles, are exposed to more dating violence than men. Women may even internalize the violence to which society exposes them and turn it into misogyny towards their fellow men.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be over 18 years of age
* The participant is a woman
* The participant's ability to read, speak and write Turkish
* The participant must have had a dating relationship at least once in his or her life or is currently in a dating relationship.

Exclusion Criteria:

* Students who agree to participate in the research but do not attend any sessions of the training, who do not want to fill out the required surveys at any stage of the research, or who want to withdraw from the research at any stage of the research will be excluded from the sample.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female students were preferred to study dating violence against women and internalized misogyny.
Enrollment: 48 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2024-01-10 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
The impact of Peer Education Based on Assertiveness Skills | Within 2 month
  The behavioral change attitude that occurs 1 week after the training will be measured according to the Passivity, Assertiveness and Aggression Scale, Internalized Misogyny Scale and Dating Violence Attitude Scale scores.
  Passivity, Assertiveness and Aggression Scale: Total score varies between 10 and 40. While low scores from the scale indicate high levels of passivity, assertiveness and aggression, high scores indicate low levels of passivity, assertiveness and aggression.
  Internalized Misogyny Scale: The total score that can be obtained from the scale varies between 17-119, and as the score increases, internalized misogyny also increases.
  Dating Violence Attitude Scale: The highest score that can be obtained from each item is 5 and the lowest score is 1. The average score of the scale approaching 5 indicates that individuals' attitudes towards dating violence are negative and they do not support dating violence behaviour.

IPD SHARING:
Plan to Share IPD: No